CLINICAL TRIAL: NCT05136664
Title: A 2-Part, Single-Blind, Phase 3 Trial Evaluating the Efficacy and Safety of Patiromer for the Treatment of Hyperkalaemia in Chinese Subjects (The Patiromer JADE Study)
Brief Title: Trial Evaluating the Efficacy and Safety of Patiromer in Chinese Subjects
Acronym: Patiromer JADE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vifor Fresenius Medical Care Renal Pharma (Industry)
Collaborators: Tigermed Consulting Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PAT-CHINA-303; CTR20212173 (Registry Identifier: Center for Drug Evaluation (CDE), NMPA)
Record Dates: First submitted 2021-11-15; First posted 2021-11-29 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Hyperkalemia; Renal Insufficiency, Chronic
Keywords: Hyperkalemia; Chronic kidney disease
MeSH Terms: conditions — Hyperkalemia; Renal Insufficiency, Chronic | interventions — Suspensions

STUDY DESIGN:
Intervention Model Description: 2-part, single-blind, randomised withdrawal, placebo-controlled (Part B), parallel group study that includes a 4-week patiromer treatment phase (Part A) followed by an 8-week randomised placebo-controlled withdrawal phase (Part B).
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part A: Patiromer (Experimental): Part A: 4-week, single-arm patiromer treatment phase (4 weeks)
  Interventions: Drug: Patiromer Powder for Oral Suspension (Part A)
- Part B: Placebo (Placebo Comparator): Part B: 8-week randomized, parallel group, placebo-controlled withdrawal phase
  Interventions: Drug: Placebo (Part B)
- Part B: Patiromer (Experimental): Part B: 8-week randomized, parallel group, placebo-controlled withdrawal phase
  Interventions: Drug: Patiromer Powder for Orals Suspension (Part B)

INTERVENTIONS:
Drug: Patiromer Powder for Oral Suspension (Part A) — Participants initiate patiromer at an oral dose of 1 packet/day (8.4g/day as powder for suspension). The dose is adjusted ate the following visit based on local serum potassium (sK+) levels.
  The content of each packet should be mixed with water, apple or cranberry juice before administration.
  Arms: Part A: Patiromer
Drug: Placebo (Part B) — Placebo is provided in packets, each containing 6 g of placebo as powder for suspension. Participants will take 1 packet per day, by mixing its content with water, apple or cranberry juice.
  Arms: Part B: Placebo
Drug: Patiromer Powder for Orals Suspension (Part B) — Participants will continue to receive the same number of packets established during Part A, but dose may be up- or down titrated depending on sK+ levels.
  The content of each packet should be mixed with water, apple or cranberry juice before administration.
  Arms: Part B: Patiromer

SUMMARY:
This is a multicentre, 2-part, single-blind, randomised, withdrawal, placebo-controlled study, that includes a 4-week patiromer treatment phase (Part A) followed by an 8-week randomised placebo-controlled withdrawal phase (Part B) and a 2-week follow-up period.

DETAILED DESCRIPTION:
In Part A, participants who meet all eligibility criteria will initiate patiromer at an oral dose of 8.4 g (1 packet/day). The dose will be adjusted based on the serum potassium (sK+) levels.

After the completion of part A, all the participants who meet the eligibility criteria for Part B will be randomised to receive patiromer or placebo. Participants will start Part B with the same dose of patiromer they were receiving at the end Part A. However, Patiromer dose may be up- or down-titrated based on sK+ levels.

The primary objectives of the study are:

Part A - To evaluate the efficacy of patiromer for the treatment of hyperkalemia in Chinese subjects.

Part B - To evaluate the effect of withdrawing patiromer on sK+ control. To determine if the treatment with patiromer will result in continued use of renin-angiotensin-aldosterone system inhibitor (RAASi) medications.

ELIGIBILITY:
Inclusion Criteria:

* - Chinese subjects at least 18 years of age.
* - Chronic Kidney Disease (CKD) stage 3 and 4.
* - Mean of 2 measurement of serum potassium higher than 5.0 and lower than 6.5 mEq/L at baseline.
* - Subjects on any stable dose of at least 1 RAASi medication for at least 28 days before Day 0/baseline.
* - If on antihypertensive medication, have a stable dose for 28 days before Day 0/baseline.
* - Women of childbearing potential must agree to continue using contraception throughout the study and for 4 weeks after study completion.

Exclusion Criteria:

* - Any level of hyperkalemia at Day 0/baseline that, in the opinion of the Investigator, requires emergency intervention.
* - Type 1 diabetes or Type 2 diabetes mellitus with glycated haemoglobin (Hb A1c) higher than 10.0% at screening/Part A baseline.
* - History of acute renal insufficiency in the past 3 months prior to the beginning of the study.
* - Diseases affecting the hearth muscle and heart's ability to pump blood around the body
* - Major surgery including thoracic and cardiac within 3 months prior to the beginning of the study or anticipated need during study participation.
* - Heart or kidney transplant recipient or anticipated need for transplant during study participation
* - Diagnosis or treatment of a malignancy in the past 2 years before Day 0/baseline.
* - Use of potassium supplements, bicarbonate or baking soda in the last 7 days prior to Day 0/baseline.
* - Pregnant women or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2022-02-10 (Actual); Primary Completion 2025-11-18 (Actual); Study Completion 2025-11-18 (Actual)

PRIMARY OUTCOMES:
Part A: Change from baseline in the serum potassium (sK+) | Week 4
  Measured in milliequivalents per litre (mEq/L)
Part B: Change from Week 4 in sK+ | The earlier of: Week 8 or the date when RAASi therapy is first decreased or discontinued
  Measured in mEq/L

SECONDARY OUTCOMES:
Part A: Proportion of participants having an sK+ level between 3.8 and less than 5.1 mEq/L at Week 4 | Week 4
Part B: Proportion of participants taking any RAASi medication at Week 12 | Week 12
Part B: Proportion of subjects discontinuing/reducing RAASi medication due to hyperkalemia | From Week 4 to 2 weeks after the end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Julian Platon, MD, PhD, Study Director — CSL Vifor
Locations (29):
- China (29):
  - Investigator Site 009, Hefei, Anhui
  - Investigator Site 008, Hefei, Anhui
  - Investigator Site 016, Beijing, Beijing Municipality
  - Investigator Site 012, Lanzhou, Gansu
  - Investigator Site 003, Lanzhou, Gansu
  - Investigator Site 029, Guangzhou, Guangdong
  - Investigator Site 030, Nanning, Guangxi
  - Investigator Site 024, Nanyang, Henan
  - Investigator Site 010, Wuhan, Hubei
  - Investigator Site 006, Changsha, Hunan
  - Investigator Site 002, Changzhou, Jiangsu
  - Investigator Site 019, Nanjing, Jiangsu
  - Investigator Site 021, Wuxi, Jiangsu
  - Investigator Site 005, Xuzhou, Jiangsu
  - Investigator Site 013, Zhenjiang, Jiangsu
  - Investigator Site 007, Changchun, Jilin
  - Investigator Site 018, Yinchuan, Ningxia
  - Investigator Site 028, Shanghai, Pudong New Area
  - Investigator Site 015, Shanghai, Shanghai Municipality
  - Investigator Site 022, Taiyuan, Shanxi
  - Investigator Site 011, Yuncheng, Shanxi
  - Investigator Site 004, Chengdu, Sichuan
  - Investigator Site 014, Tianjin, Tianjin Municipality
  - Investigator Site 027, Zhuzhou, Tianyuan District
  - Investigator Site 023, Ürümqi, Xinjiang
  - Investigator Site 001, Hangzhou, Zhejiang
  - Investigator Site 020, Hanzhou, Zhejiang
  - Investigator Site 026, Jiaxing, Zhejiang
  - Investigator Site 025, Jinhua, Zhejiang

IPD SHARING:
Plan to Share IPD: No